CLINICAL TRIAL: NCT04394767
Title: Couple and Spouse Caregiver in Huntington's Disease
Acronym: COCOON
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision, no more inclusions made since the last extension
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_33; 2018-A02046-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-10-16; First posted 2020-05-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; spouse caregiver; quality of life
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives are to better document the psychosocial status and needs of caregiver of HD patients and understand the dyad functioning, facing the disease at various stages.

ELIGIBILITY:
Inclusion Criteria:

For patient :

* HD, CAG > 36, motor UHDRS > 5
* Being able to communicate with the investigator

For both spouses :

* Living together since at least 5 years
* 30 to 60 years old

Exclusion Criteria:

For patient :

- Other chronic neurologic disorder

For both spouses :

* Psychiatric disease
* Unable to participate, incl read, understand and sign the informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Huntington disease population ( patient, caregiver, spouses)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
report of the experience and interactions of couple and Spouse Caregiver in Huntington's Disease | once time, Baseline
  Qualitative assessment: Interpretative phenomenological analysis (IPA) by semi-structured interviews to explore families representations and strategies about the patients with Huntington's Disease

SECONDARY OUTCOMES:
report of the experience and interactions of couple and Spouse Caregiver in Huntington's Disease | once time, Baseline
  Qualitative assessment : Thematic analysis by COAT (Carers Outcome Agreement Tool) during a semi-structured interviews to explore families representations and strategies about the patients with Huntington's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Clémence Simonin, MD, Principal Investigator — University Hospital, Lille; Pascal ANTOINE, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU Lille, Lille, France